CLINICAL TRIAL: NCT03830359
Title: Efficacy and Safety Assessment of T2769 in Patients With Moderate to Severe Dry Eye Syndrome
Brief Title: Efficacy, Safety of T2769 in Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LT2769-001
Record Dates: First submitted 2019-01-07; First posted 2019-02-05 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T2769 (Experimental): T2769 Ophthalmic solution patients treated with 1 drop in each eye 3 to 6 times daily
  Interventions: Other: T2769

INTERVENTIONS:
Other: T2769 — At least 55 enrolled patients for at least 50 evaluable patients treated by T2769 for 42 days
  Other Names: Ophthalmic solution

SUMMARY:
Efficacy of T2769 in Dry Eye Desease

DETAILED DESCRIPTION:
Multicenter and open study

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Male or female aged from ≥ 18 years old
* Known Dry Eye Syndrome requiring artificial tears within the last 3 months prior to study screening

Exclusion Criteria:

* Best far corrected visual acuity ≤ 2/10
* Severe blepharitis Severe dry eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lamia El Fekih, Pr, Principal Investigator — fekihlamia63@gmail.com
Locations (3):
- Tunisia (3):
  - Hôpital Universitaire Tahar Sfar, Mahdia
  - "Hôpital Universitaire Fattouma Bourguiba, Monastir
  - "Hôpital de Forces de Sécurité Intérieure La Marsa, Tunis

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- T2769: T2769 : 1 drop in each eye 3 to 6 times daily during 42 days
Period: Overall Study
Arm/Group | T2769
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- T2769: T2769 Ophthalmic solution One drop in each eye 3 to 6 times daily
  T2769: 62 patients treated by T2769 for 42 days
Arm/Group | T2769
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 62
Region of Enrollment [Number; unit: participants]
  Tunisia | 62

OUTCOME MEASURES:

1. Primary Outcome: Ocular Symptomatology
Description: Change from baseline in ocular symptomatology on a Visual Analog Scale (0=No discomfort and 100=Maximal discomfort) at Day 42.
Time Frame: Baseline and Day 42
Population: m-ITT population : all enrolled patients having received at least one dose of the IP and with at least one baseline and post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | T2769
Number analyzed (Participants) | 62
units on a scale | -55.9 (23.1)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- T2769: T2769 Ophthalmic solution One drop in each eye 3 to 6 times daily of T2769 for 42 days
Arm/Group | T2769
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03830359/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT03830359/SAP_001.pdf